CLINICAL TRIAL: NCT02179112
Title: Determining Universal Processes Related to Best Outcome in Emergency Gastrointestinal Surgery: an International Evaluation
Acronym: GlobalSurg-1
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: NR/1404AB12
Record Dates: First submitted 2014-06-29; First posted 2014-07-01 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2021-06

CONDITIONS: Surgical Procedures, Operative
Keywords: Surgery; Specialties, Surgical; Geography, Medical; Developing Countries; Developed Countries; Laparotomy; Outcome and Process Assessment (Health Care); Treatment Outcome; Quality of Health Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Emergency Abdominal Surgery — Emergency intra-peritoneal surgery (only exclusion: Caesarian section).

SUMMARY:
A multicentre, international evaluation of emergency abdominal surgery to establish surgical outcomes and identify common, modifiable best practice processes.

DETAILED DESCRIPTION:
Background: With over 200 million surgical operations per year worldwide and with nearly every acute hospital providing surgical services, outcomes from emergency general surgery represent internationally important healthcare markers. Best practice and modifiable processes that are relevant to good patient outcomes around the world require validation using patient-level data.

Aim: The primary aim of this study is to identify internationally relevant, modifiable surgical practices (in terms of modifiable equipment and clinical management) associated with best care. These factors will include use of imaging, supplementary oxygen, pulse oximetry, critical care, and safety checklists.

Method: This is a multicentre, international, prospective cohort study. Any hospital in the world performing acute surgery will be eligible to enter. Any patient undergoing emergency surgery with an incision entering the peritoneal cavity is eligible. Routine, anonymised clinical data on consecutive patients will be collected over a two week period in each surgical centre, with up to 30 days follow-up data collected. The primary outcome is 24-hour post-operative mortality rate. Secondary outcomes include 30-day inpatient post-operative mortality rate, and 30-day serious complication rate. Participating centres will also be asked to complete a survey that will collect data on hospital structural and resource characteristics.

Data will be entered and stored securely via the University of Edinburgh's REDCap system. This pragmatic protocol (which will delivered across many low-resource settings) does not allow for independent verification of data entry. Data collection norms are laid out in the protocol, where data definitions are also clearly provided. Sample size is not relevant to this exploratory audit. Centres will only be included where there is at least 95% data completeness.

Potential explanatory variables that will be explored in subsequent analysis include country Human Developmental Index, and resource differences.

ELIGIBILITY:
Centre Inclusion Criteria:

* Any acute surgical unit worldwide is eligible to enter
* All participating centres will be required to register their details, complete an online training module, and complete a pilot audit prior to commencing.
* Centres must ensure that they can include consecutive patients and provide at least 95% data completeness.
* There is no minimum number of patients per centre, as long as the patient(s) included are consecutive.

Inclusion Criteria:

* All sequential patients undergoing emergency intra-peritoneal surgery during the chosen 2-week period should be included.
* Emergency (unplanned, non-elective, same admission) procedures only. This includes patients undergoing an emergency re-operation after a previous procedure on the same in-patient stay.
* Laparoscopic, laparoscopic converted and open cases can be included.
* Any age patient (adult and paediatric) can be included.

Exclusion Criteria:

* Elective (planned) or semi-elective (where patient initially admitted as an emergency, then discharged from hospital, and re-admitted at later time for surgery) procedures.
* Caesarean section. These patients represent a separate operative group, with different priorities and treatment pathways. They have been studied in detailed elsewhere, and their frequency would skew the results of this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from all acute surgical units worldwide which provide an emergency surgery service.
Sampling Method: Probability Sample
Enrollment: 10745 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
24-hour peri-operative mortality rate | At 24 hours following conclusion of the operation
  Number of deaths during operation or within 24 hours of operation conclusion, divided by number of operations undertaken.

SECONDARY OUTCOMES:
30-day peri-operative mortality rate (POMR-30) | Up to 30 days from the operation (or point of discharge- see definition)
  Number of deaths during operation or within 30 days of operation, or at the point of final discharge if out-patient mortality status unknown.
  Please see reference for justification of our use of this definition in our global cohort.
  - - -
  Watters DA, Hollands MJ, Gruen RL, Maoate K, Perndt H, McDougall RJ, et al. Perioperative Mortality Rate (POMR): A Global Indicator of Access to Safe Surgery and Anaesthesia. World J Surg. 2014 May 20;1-9.
30-day peri-operative serious complication rate | Up to 30 days from the operation (or point of final discharge - see below)
  Number of serious complications occurring, divided by number of operations. Measured at operation or within 30 days of operation, or point of final discharge if out-patient information unavailable. (See definition of POMR-30 above for justification).
  Serious complications defined as Grade III or V within the Clavien-Dindo classification (Grade III = complications requiring surgical, endoscopic or radiological intervention; Grade V = death).
  - - -
  Dindo D, Demartines N, Clavien P-A. Classification of Surgical Complications. Ann Surg. 2004 Aug;240(2):205-13.

CONTACTS AND LOCATIONS:
Overall Officials: Ewen M Harrison, PhD, FRCS, Principal Investigator — University of Edinburgh; Aneel Bhangu, MBChB, MRCS, Study Director — University of Birmingham; J E Fitzgerald, BA, MRCS, Study Director — Lifebox Foundation; Stuart J Fergusson, BSc, MRCS, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Result] GlobalSurg Collaborative. Laparoscopy in management of appendicitis in high-, middle-, and low-income countries: a multicenter, prospective, cohort study. Surg Endosc. 2018 Aug;32(8):3450-3466. doi: 10.1007/s00464-018-6064-9. Epub 2018 Apr 5. PMID 29623470
- [Derived] GlobalSurg Collaborative. Determinants of morbidity and mortality following emergency abdominal surgery in children in low-income and middle-income countries. BMJ Glob Health. 2016 Dec 12;1(4):e000091. doi: 10.1136/bmjgh-2016-000091. eCollection 2016. PMID 28588977
- [Derived] GlobalSurg Collaborative. Mortality of emergency abdominal surgery in high-, middle- and low-income countries. Br J Surg. 2016 Jul;103(8):971-988. doi: 10.1002/bjs.10151. Epub 2016 May 4. PMID 27145169
- [Derived] Bhangu A, Fitzgerald JE, Fergusson S, Khatri C, Holmer H, Soreide K, Harrison EM. Determining universal processes related to best outcome in emergency abdominal surgery: a multicentre, international, prospective cohort study. BMJ Open. 2014 Oct 29;4(10):e006239. doi: 10.1136/bmjopen-2014-006239. PMID 25354824
- See also: Full protocol - online — http://globalsurg.org/protocol/